CLINICAL TRIAL: NCT04957810
Title: Evaluation of the Effect of Using WeChat Applet to Intervene in the Home Functional Exercise of Patients After Anterior Cruciate Ligament Reconstruction Based on the Health Belief Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: M2019069
Record Dates: First submitted 2021-06-25; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients who are given regular home functional exercises and discharged from the hospital (No Intervention): Discharge guidance using regular home function exercises, that is, existing regular missions and paper-based brochures
- Patients who are guided by conventional discharge guidance and the optimized WeChat official account (Active Comparator): Use regular discharge guidance and optimized WeChat public account guidance
  Interventions: Behavioral: WeChat Mini Program

INTERVENTIONS:
Behavioral: WeChat Mini Program — Through the WeChat applet, it provides services such as visit content configuration, self-image configuration, self-image measurement configuration, and visit reminders.
  Arms: Patients who are guided by conventional discharge guidance and the optimized WeChat official account

SUMMARY:
Based on the home rehabilitation exercise of patients undergoing ACL reconstruction, the existing WeChat applet of sports medicine of the Third Hospital of Beijing Medical University is optimized to be used as a health education tool to guide patients undergoing home rehabilitation exercise after ACL reconstruction.

DETAILED DESCRIPTION:
With the development of national fitness and sports, the incidence of ACL injury is increasing year by year. ACL reconstruction is the best way to treat ACL injuries, and the success rate of the operation is high, but patients still need to recover after surgery, otherwise, it will be difficult to fully restore knee joint function. However, my country's rehabilitation medical resources are obviously insufficient. After discharge from the hospital, ACL reconstruction patients usually go home and exercise at home according to the rehabilitation plan formulated by the surgeon or rehabilitation physician. However, compliance is still poor, and rehabilitation is relatively difficult to achieve the expected results, which affects the lives of patients quality. The WeChat official account and its affiliated mini-programs have been widely used in different health fields as a means of health communication. The health belief model is a guiding theory commonly used in the field of health education to guide patients to make behavior changes. This study intends to use the functional advantages of the WeChat applet to explore the optimization of the existing Peking University Third Hospital Sports Medicine WeChat applet based on the health belief model and to use the postoperative rehabilitation of patients undergoing ACL injury reconstruction as a pilot to evaluate the optimized The WeChat Mini Program can improve the intervention effect of patients' home functional exercise compliance after ACL injury reconstruction, to provide effective health education for more extensive sports medicine-related home functional exercises, improve their rehabilitation effects and quality of life, and better To ensure the efficacy of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 years old (including 18 years old) and 45 years old;
2. Patients who underwent simple ACL reconstruction for the first time, combined with cartilage trimming and partial meniscus resection, and had the same postoperative rehabilitation plan;
3. Those who have basic literacy and communication skills;
4. Those who have a smartphone, can use WeChat or can learn to use WeChat;

Exclusion Criteria:

1. Have a history of joint infection, joint tuberculosis or osteomyelitis, or have undergone surgery in the lower limbs within 6 months;
2. Combined with severe heart, brain, kidney, and other organ dysfunction;
3. Patients with other severe knee joint disease injuries;
4. The patient is accompanied by mental illness or cognitive impairment, unable to study and participate in rehabilitation training;
5. Those who have participated in other similar rehabilitation function training programs, or transferred to other medical institutions for rehabilitation after being discharged from the hospital;
6. Those who have not signed the informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in range of motion of knee joint | 2 weeks, 6 weeks and 12 weeks after surgery
  Changes in range of motion of the knee between two time points

SECONDARY OUTCOMES:
Visual pain score during knee motion angle exercise | 2 weeks, 6 weeks and 12 weeks after surgery
  Visual pain score during knee motion angle exercise were measured at 2,6 and 12 weeks.
SF-12 quality of life scale | 2 weeks, 6 weeks and 12 weeks after surgery
  SF-12 means the 12-items Short Form Health Survey.Patients' scores were measured at 2,6 and 12 weeks ,and the higher the score ,the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: yuping yang, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No